CLINICAL TRIAL: NCT03631615
Title: A Phase II Study of Neoadjuvant Chemoradiation Plus PD-1 Antibody(SHR-1210) in the Locally Advanced Proximal Stomach Adenocarcinoma (Neo-PLANET)
Brief Title: Neoadjuvant Chemoradiation Plus PD-1 Antibody(SHR-1210) in Locally Advanced Proximal Stomach Adenocarcinoma
Acronym: Neo-PLANET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Tianshu Liu, Director of Oncology Department, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-CRT-GC-IIT
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Gastric Adenocarcinoma
Keywords: neoadjuvant chemoradiation; PD-1 antibody(SHR-1210); locally advanced proximal stomach adenocarcinoma
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therpy (Experimental): neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210)
  Interventions: Drug: Neoadjuvant chemoradiation plus PD-1 antibody(SHR-1210)

INTERVENTIONS:
Drug: Neoadjuvant chemoradiation plus PD-1 antibody(SHR-1210) — Patients will be given the perioperative treatment as below once recruited:
  1. induction Neochemotherapy (3w): one cycle of XELOX regimen before surgery;
  2. within one week after the induction, concurrent neochemoradiation will be started (5w): intensity modulated radiotherapy was given for tumors and high-risk lymphatic drainage areas.
  3. consolidation neochemotherapy will be started in 2-3w after concurrent chemoradiation: one cycle of XELOX regimen; From the beginning of induction chemo to 3w before surgery, PD-1 antibody SHR-1210 will be given q3W.
  Re-evaluation will be conducted in 1-3w after consolidation chemo, resectable patients will receive D2 resection.
  Adjuvant chemo: We advise starting 4 cycles of XELOX regimen in 4-6w after surgery.
  Other Names: Newplan

SUMMARY:
1. Target population: patients with resectable locally advanced proximal (including gastroesophageal junction, fundus and upper body) stomach adenocarcinoma (cT3-4aN+M0).
2. Primary objective: pathological complete remission (pCR) rate of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210) in patients with locally advanced proximal stomach adenocarcinoma.

Secondary objectives:

1. pathological remission rate (pRR) of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210)
2. objective response rate (ORR) of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210)
3. progression free survival (PFS)/ overall survival (OS) of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210)
4. safety of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210)

3.Trial design: This is a monocenter, single arm, phase II study to evaluate the efficacy and safety of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210) in patients with locally advanced proximal stomach adenocarcinoma.

4.Treatment plan:

Patients will be given the perioperative treatment as below once recruited:

1. induction chemotherapy (3w): one cycle of XELOX regimen (capecitabine 1000 mg/m2 bid*14d + oxaliplatin 130mg/m2, d1, Q21d);
2. within one week after the induction, concurrent chemoradiation will be started (5w): intensity modulated radiotherapy was given for tumors and high-risk lymphatic drainage areas, total dose:45Gy/25d, 1.8Gy/d, capecitabine (850 mg/m2, bid, po) will be given during radiotherapy as sensitizer.
3. consolidation chemotherapy will be started in 2-3w after concurrent chemoradiation: one cycle of XELOX regimen (capecitabine 1000 mg/m2 bid*14d + oxaliplatin 130mg/m2, d1, Q21d); From the beginning of induction chemo to 3w before surgery, PD-1 antibody SHR-1210 will be given（200mg, iv, q3w).

Re-evaluation will be conducted in 1-3w after consolidation chemo, resectable patients will receive D2 resection.

Adjuvant chemo: We advice starting 4 cycles of XELOX regimen (capecitabine 1000 mg/m2 bid*14d + oxaliplatin 130mg/m2, d1, Q21d) in 4-6w after surgery.

5.Number of subjects: 36 patients. Number of centers: 1 sites ( Fudan University Affiliated Zhongshan Hospital, which has high volume of gastric operations in China, more than 500 per year).

DETAILED DESCRIPTION:
Backgrounds:

SHR-1210 is a PD-1 antibody developed by Jiangsu Heng Rui Medicine Co. Nowadays, fifteen clinical trials of this drug have been conducted in patients with different types of advanced malignant tumor, including one combined with radiotherapy and three combined with chemotherapy. Until now, SHR-1210 has exhibited favorable safety in recruited patients. Incidence rate of SAE is only 1%.

Several big scale clinical research like POET, RTOG 9904 and TOPGEAR have proofed the efficacy and safety of neoadjuvant chemoradiation in treating locally advanced GEJ cancer or gastric cancer.

Study design:

This clinical trial will be conducted under Simon's optimal two-stage design. The first stage needs 15 participants, if ≥1 participants acquire remission, then the study will move on to the second stage and enroll the rest 21 participants. The total sample size will be 36 patients.

We will shut down the study in advance, if situations below happens: 1) 1 treatment related death, >3 disease progression or >2 hyper-progressive disease happen during the first stage; 2) 2 treatment related death, >6 disease progression or >4 hyper-progressive disease happen during the whole study.

Patients with abnormal autoimmune status, unfavorable body function, factors impeding drug taking, absorption and metabolism will be excluded. Study participants with disease progression or severe/ intolerant toxicity during treatment will withdraw the study.

Hyper-progressive disease is defined as 1) progression 2) more than doubled growth rate 3) tumor volume increase >50% in 2 months after initialing the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. histologically documented gastric adenocarcinoma.
2. primary lesion is in proximal stomach, including gastroesophageal junction, fundus and upper body.
3. clinically diagnosed stage T3-4aN+M0 according to ultrasound endoscopy or enhanced CT/MRI scan.
4. at least one evaluable lesion in abdominal CT/MRI according to RESIST 1.1 is required.
5. surgeons participating in this study consider the lesion a resectable one.
6. Karnofsky score≥ 80.
7. Physical condition and adequate organ function to ensure the success of abdominal surgery.
8. Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥90g/L.
9. Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN in the absence of liver metastases, or < 5 × ULN in case of liver metastases. ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L.
10. Adequate renal function: Serum creatinine ≤ 1.5 x ULN, and creatinine clearance ≥ 60 ml/min.
11. Adequate coagulation function: INR/PT≤ 1.5 x ULN, aPTT≤ 1.5 x ULN.
12. No serious concomitant disease that will threaten the survival of patients to less than 5 years.
13. Male or female. Age ≥ 18 years and ≤75 years.
14. Written (signed) informed consent.
15. Good compliance with the study procedures, including lab and auxiliary examination and treatment.
16. Female patients should not be pregnant or breast feeding.
17. Agree to take contraception measures during treatment and in 120 days after last dose of SHR-1210 or in 180 days after last dose of chemo.

Exclusion Criteria:

1. patients with distant metastasis or unresectable primary lesion.
2. patients with T1, T2 lesion according to CT/MRI or ultrasound endoscopy.
3. history of chemo, radiation, immune therapy or radical resection for the stomach adenocarcinoma, except steroids.
4. patients with active autoimmune disease or history of refractory autoimmune disease.
5. patients with active malignant tumor in recent 2 years, except the tumor studied in this research or cured locally tumor like resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ.
6. uncontrollable pleural effusion, pericardial effusion, or ascites in 2 weeks before recruitment.
7. patients who have digestive tract bleeding in 2 weeks before recruitment or with high risk of bleeding.
8. perforation / fistula of GI tract in 6 months before recruitment.
9. patients with upper GI tract obstruction or functional abnormality or malabsorption syndrome, which can affect absorption of capecitabine.
10. losing over 20% body weight in 2 months before recruitment.
11. pulmonary disease history: interstitial pulmonary disease, non-infective pneumonitis, pulmonary fibrosis, acute pulmonary disease.
12. uncontrollable systemic diseases, including diabetes, hypertension, etc.
13. severe chronic or active infections in need of systemic antibacterial, antifungal, or antiviral treatment, including TB or HIV, etc.
14. patients with untreated chronic hepatitis B or HBV DNA over 500 IU/ml or positive HCV RNA.
15. patients with any cardiovascular risk factors below:

    1. cardiac chest pain occurring in 28 days before recruitment, defined as moderate pain that limits daily activity.
    2. pulmonary embolism with symptoms occurring in 28 days before recruitment.
    3. acute myocardial infarction occurring in 6 months before recruitment.
    4. any history of heart failure reaching grade 3/4 of NYHA in 6 months before recruitment.
    5. ventricular arrhythmias of Grade 2 or grater in 6 months before recruitment, or accompanied by supraventricular tachyarrhythmias requiring medical treatment.
    6. cerebrovascular accident within 6 months before recruitment.
16. patients with peripheral neuropathy NCI CTC AE grade 1, except those with only deep tendon reflex disappearing.
17. moderate or severe renal injury [creatinine clearance rate≤50 ml/min (according to Cockroft & Gault equation)], or Scr>ULN.
18. dipyrimidine dehydrogenase (DPD) deficiency.
19. allergic to any drug in this study.
20. history of allogeneic stem cell transplantation or organ transplantation.
21. use of steroids (dosage>10mg/d prednisone) or other systemic immune suppressive therapy in 14 days before recruitment, except patients treated with regimens below: a. steroids for hormone replacement (dosage>10mg/d prednisone); b. steroids for local application with little systemic absorption; c. short -term (≤ 7 days) steroids for preventing allergy or vomiting.
22. vaccinated with live vaccine in 4 weeks before recruitment.
23. receiving immune (interleukin, interferon, thymin) treatment or treatment of other trials in 28 days before recruitment.
24. receiving palliative radiation in 14 days before recruitment.
25. history of anti PD-1, PD-L1, PD-L2 or any other specific T cell co-stimulation or checkpoint pathway targeted treatment.
26. receiving operation in 28 days before recruitment, only if the operation is a minimally invasive one e.g. PICC.
27. for patients with uncontrolled epilepsy, CNS diseases or history of mental disorder, researchers should evaluate whether their diseases will impede their signing of informed consent or compliance of treatment.
28. existing of potential situation which will impede drug administration or affect toxicity analysis or alcohol/ drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete remission (pCR) rate of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210) in patients with locally advanced proximal stomach adenocarcinoma. | 5 months after the last subject participating in
  rate of patients with no residual tumor lesion (Grade 3) in surgical specimen

SECONDARY OUTCOMES:
pathological remission rate (pRR) of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210) | 5 months after the last subject participating in
  rate of patients with < 2/3 residual tumor lesion (Grade 1b, 2, 3) in surgical specimen compared to baseline
objective response rate (ORR) of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210) | 36 months after the last subject participating in
  rate of patients with complete remission (CR) or partial remission (PR) based on RESIST1.1. ORR was evaluated by chest, abdominal & pelvic CT/MRI. Evaluation will be conducted on 9w&15w during preoperative treatment, every 6 weeks during adjuvant XELOX, and every 0.5 year after all treatments.
progression free survival (PFS) of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210) | 36 months after the last subject participating in
  PFS is defined as time interval from recruitment to tumor progression or censoring. Tumor progression is defined as below: 1) relapse of primary lesion 2) emerging of new lesion 3) distant metastasis 4) death of any reason 5)tumor progression according to RESIST 1.1 on CT/MRI.
overall survival (OS) of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210) | 36 months after the last subject participating in
  OS is defined as time interval from recruitment to all-caused death or censoring.
safety of neoadjuvant chemoradiation plus PD-1 antibody (SHR-1210) | 1 month after the last date of treatment
  Adverse events (AE) of chemo- and radio-therapy will be graded and documented according to NCI-CTC AE v4.03 from the beginning of treatment to 1 months after the last date of treatment. Documentary will include severity, lasting period and occurrence time. Main AEs include vomiting, diarrhea, anemia, leukopenia, thrombocytopenia, hand-foot syndrome, epidermal capillary hyperplasia, immune related adverse events (including pneumonia, interstitial lung disease, AST/ALT elevations, rash, diarrhea, hypothyroidism and hyperthyroidism) and hyper-progressive tumor.
  AEs of surgery refer to complications which happen during or in 30 days after operation. Severe complications after operation such as abdominal or GI tract bleeding, anastomotic fistula, pancreatic fistula of grade B or above, incision complications (infection, bleeding, rupture) will be observed and classified by Clavien-Dindo grading.

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Doctor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China